CLINICAL TRIAL: NCT00375674
Title: Sunitinib Treatment Of Renal Adjuvant Cancer (S-trac): A Randomized Double-blind Phase 3 Study Of Adjuvant Sunitinib Vs. Placebo In Subjects At High Risk Of Recurrent Rcc
Brief Title: A Clinical Trial Comparing Efficacy And Safety Of Sunitinib Versus Placebo For TheTreatment Of Patients At High Risk Of Recurrent Renal Cell Cancer
Acronym: S-TRAC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A6181109; 2006-004024-37 (EudraCT Number); S-TRAC (Other: Alias Study Number)
Record Dates: First submitted 2006-09-12; First posted 2006-09-13 (Estimated); Results first posted 2017-08-18 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-08

CONDITIONS: Kidney Neoplasms
MeSH Terms: conditions — Kidney Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: Sunitinib malate
- B (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sunitinib malate — sunitinib malate 50 mg PO on schedule 4/2: 4 weeks on, 2 weeks off for 1 year or until disease recurrence or occurrence of a secondary malignancy, significant toxicity, or withdrawal of consent.
  Arms: A
Other: Placebo — Placebo PO for 1 year on schedule 4/2: 4 weeks on, 2 weeks off or until disease recurrence or occurrence of a secondary malignancy, significant toxicity, or withdrawal of consent
  Arms: B

SUMMARY:
To compare the disease free survival time and safety of sunitinib with placebo in adjuvant treatment patients at high risk of recurrent kidney cancer after surgery.

ELIGIBILITY:
Inclusion Criteria:

* High risk renal cancer per modified UISS criteria
* Eastern Cooperative Oncology Group (ECOG) 0-2
* predominant clear cell histology
* No prior anti-cancer treatment
* Kidney tumor has been removed
* No evidence of macroscopic disease following surgery

Exclusion Criteria:

* Histologically undifferentiated carcinomas or collecting duct carcinoma, lymphoma, sarcoma or subjects with metastatic renal sites.
* Diagnosis of any second malignancy within the last 5 years, except basal cell carcinoma, squamous cell skin cancer, or in situ carcinoma of the cervix uteri that has been adequately treated with no evidence of recurrent disease for 12 months
* known HIV or Hepatitis
* any severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 674 (Actual)
Dates: Start 2007-08-01 (Actual); Primary Completion 2016-04-07 (Actual); Study Completion 2017-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (114):
- United States (12):
  - Ronald Reagan UCLA Medical Center Department of Pharmaceutical Services, Los Angeles, California
  - UCLA Clark Urology Center, Los Angeles, California
  - Emory University Hospital, Atlanta, Georgia
  - The Emory Clinic, Inc, Atlanta, Georgia
  - Hematology and Oncology Specialists, LLC, Marrero, Louisiana
  - Hematology and Oncology Specialists, LLC, Metairie, Louisiana
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Intermountain Medical Center, Murray, Utah
- Monash Medical Centre - Moorabin Campus, East Bentleigh, Victoria, Australia
- China (13):
  - Urology Department, Sun Yet-Sen University Cancer Center, Guangzhou, Guangdong
  - The first affiliated hospital of Soochow university/Department of Urology, Suzhou, Jiangsu
  - Fudan University Cancer Hospital, Department of Urology, Shanghai, Shanghai Municipality
  - Urology Department, Renji Hospital,Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Department of Urology, Shanghai Changhai Hospital, Shanghai, Shanghai Municipality
  - Department of Urology, the Second Affiliated Hospital of Zhejiang University College of Medicine, Hangzhou, Zhejiang
  - Cancer Institute & Hospital, CAMS, Beijing
  - Department of Urology,Peking University First Hospital, Beijing
  - Chinese PLA General Hospital/Urology Department, Beijing
  - Urology Department, South-Western Hospital, 3rd Military Medical University., Chongqing
  - Huashan Hospital Fudan University, Shanghai
  - Tianjin Oncology Hospital, urology department, Tianjin
  - The Second Hospital of Tianjin Medical University, Tianjin
- Instituto Nacional de Cancerologia - ESE, Bogota, Cundinamarca, Colombia
- Czechia (5):
  - Masarykuv onkologicky ustav, Brno
  - Fakultni nemocnice v Motole, Klinika zobrazovacich metod, Prague
  - Fakultni nemocnice v Motole, Radioterapeuticko-onkologicke oddeleni, Prague
  - Fakultni nemocnice v Motole, Ustav nuklearni mediciny, Prague
  - Krajska zdravotni a. s., Masarykova nemocnice v Usti nad Labem, o. z., Ústí nad Labem
- Aarhus Universitetshospital, Aarhus C, Denmark
- France (11):
  - Hopital Saint-Andre, Bordeaux
  - Centre Oscar Lambret, Lille
  - Institut Paoli-Calmettes, Marseille
  - CRLC Val d'Aurelle, Montpellier
  - Hopital Europeen Georges Pompidou, Paris
  - Centre Eugene Marquis, Rennes
  - Institut de Cancerologie de l'Ouest - Centre Rene Gauducheau, Saint-Herblain
  - Hopital Civil, Strasbourg
  - Institut Claudius Regaud - Centre de Lutte Contre le Cancer, Toulouse
  - CHRU de Tours - Hopital Bretonneau, Tours
  - Institut Gustave Roussy / Service d'Immunotherapie, Villejuif
- Germany (16):
  - RWTH Aachen, Urologische Klinik, Aachen
  - Charite Universitaetsmedizin Berlin, Campus Charite Mitte, Berlin
  - Charite Universitaetsmedizin Berlin, Campus Benjamin Franklin, Berlin
  - Universitaetsklinikum Bonn, Klinik und Poliklinik fuer Urologie, Bonn
  - Universitaetsklinikum Carl Gustav Carus der Technischen Universitaet Dresden, Dresden
  - Klinikum der J. W. Goethe-Universitaet, Medizinische Klinik II, Frankfurt
  - Universitaetsklinikum Hamburg-Eppendorf, Klinik fuer Urologie, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklinikum des Saarlandes, Klinik fuer Urologie und Kinderurologie, Homburg/Saar
  - Klinikum der Friedrich-Schiller-Universitaet Jena, Universitaetsklinik und Poliklinik fuer Urologie, Jena
  - Klinik und Poliklinik fuer Urologie, UKSH Campus Luebeck, Lübeck
  - Ludwigs-Maximilians-Universitaet Muenchen, Klinikum Grosshadern Urologische Klinik und Poliklinik, München
  - Universitaetsklinikum Muenster Klinik und Poliklinik fuer Urologie, Münster
  - Klinikum Nuernberg, 5. Medizinische Klinik, Haematologie / Onkologie, Nuremberg
  - Eberhardt-Karls-Universität Tübingen, Klinik für Urologie, Tübingen
  - Universitaetsklinikum Ulm, Urologische Universitaetsklinik, Ulm
- Greece (2):
  - "Alexandra" general hospital of Athens, department of Clinical Therapeutics, Oncology Unit, Athens
  - Theageneio Anticancer Hospital, Thessaloniki
- Ireland (4):
  - AMNCH Hospital, Dublin
  - Mater Misericordiae Hospital, Dublin
  - Beaumont Hospital, Dublin
  - University Hospital Galway, Galway
- Israel (2):
  - Institute of Oncology, Davidoff Center, Petah Tikva
  - Assaf Harofeh Medical Center, Ẕerifin
- Italy (6):
  - Unita' Operativa di Oncologia Medica, Policlinico Sant'Orsola Malpighi, Bologna
  - P.O.SS. ANNUNZIATA 14° LIVELLO CORPO A, Clinica Oncologica, Chieti Scalo
  - Azienda Socio-Sanitaria Territoriale di Cremona, Ospedale di Cremona, Cremona
  - IRCCS AO Universitaria San Martino, IST Istituto Nazionale per la Ricerca sul Cancro, Genova
  - Fondazione IRCCS, Istituto Nazionale dei Tumori, SC Oncologia Medica 2, Milan
  - Divisione di Oncologia, AORN Antonio Cardarelli, Napoli
- Sarawak General Hospital, Kuching, Sarawak, Malaysia
- Torre Medica Cristobal Colon, Acapulco de Juárez, Guerrero, Mexico
- Poland (7):
  - "Vesalius" Sp. z o.o., Krakow
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej, Uniwersytecki Szpital Kliniczny nr 2 im. Wojskowej A, Lodz
  - Uniwersytecki Szpital Kliniczny nr 2 im. Wojskowej Akademii Medycznej UM-Centralny Szpital Weteranow, Lodz
  - Oddzial Chemioterapii, Szpital Kliniczny Przemienienia Panskiego Uniwersytetu Medycznego, Poznan
  - Centrum Onkologii - Instytut im. Marii Sklodowskiej-Curie, Warsaw
  - Klinika Onkologii, Wojskowy Instytut Medyczny, Warsaw
  - Klinika Urologii i Onkologii Urologicznej Akademicki Szpital Kliniczny, Wroclaw
- Slovakia (4):
  - Univerzitna nemocnica Bratislava, Bratislava
  - Narodny Onkologicky ustav, Bratislava
  - Univerzitna nemocnica Martin, Martin
  - Fakultna nemocnica s poliklinikou, Žilina
- South Korea (5):
  - Department of Internal Medicine, Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - National Cancer Center, Goyang-si, Gyeonggido, Korea, Republic of
  - Samsung Medical Center, Seoul, Korea, Republic of
  - Asan Medical Center, Seoul, Seoul Korea, Republic of
  - Korea University Anam Hospital, Seoul, Seoul Teugbyeolsi
- Spain (6):
  - Institut Catala D'Oncologia (I.C.O), L'Hospitalet de Llobregat, Barcelona
  - Complexo Hospitalario Universitario A Coruna. Hospital Teresa Herrera, A Coruña
  - Hospital Universitario Vall D'Hebron, Barcelona
  - Hospital Clinico de Barcelona, Barcelona
  - Hospital 12 de Octubre, Madrid
  - Instituto Valenciano de Oncologia, Valencia
- Sweden (6):
  - Verksamheten urologi, SU/Sahlgrenska, Gothenburg
  - Onkologiska kliniken, Universitetssjukhuset, Lund
  - Norrlands universitetssjukhus, Urologiska kliniken, Umeå
  - Akademiska sjukhuset, Uppsala
  - Urologkliniken Akademiska Sjukhuset, Uppsala
  - Centrallasarettet, Onkologkliniken, Västerås
- Switzerland (2):
  - Onkologisches Institut, Inselspital Bern, Bern
  - Kantonsspital St. Gallen, Sankt Gallen
- Taiwan (2):
  - Taichung Veterans General Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (6):
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - Ross Hall Hospital, Glasgow
  - Post Graduate Medical School, University of Surrey, Guildford
  - Guy's Hospital, London
  - St. Mary's Hospital, Imperial College, Health care NHS Trust, London
  - Medical Oncology, Patterson institute for Cancer Research, Manchester

REFERENCES:
- [Derived] Motzer RJ, Martini JF, Mu XJ, Staehler M, George DJ, Valota O, Lin X, Pandha HS, Ching KA, Ravaud A. Molecular characterization of renal cell carcinoma tumors from a phase III anti-angiogenic adjuvant therapy trial. Nat Commun. 2022 Oct 10;13(1):5959. doi: 10.1038/s41467-022-33555-8. PMID 36216827
- [Derived] Patel A, Ravaud A, Motzer RJ, Pantuck AJ, Staehler M, Escudier B, Martini JF, Lechuga M, Lin X, George DJ. Exploratory analysis of the platelet-to-lymphocyte ratio prognostic value in the adjuvant renal cell cancer setting. Future Oncol. 2021 Feb;17(4):403-409. doi: 10.2217/fon-2020-0652. Epub 2020 Oct 8. PMID 33028084
- [Derived] Ouzaid I, Kammerer-Jacquet SF, Khene Z, Ravaud A, Patard JJ, Bensalah K, Rioux-Leclercq N. Exploring Biological Predictive Factors of Progression After Surgery in High-Risk Renal Cell Carcinoma: Results From the French Cohort of the Randomized S-TRAC Trial Patients. Front Surg. 2020 Jun 5;7:26. doi: 10.3389/fsurg.2020.00026. eCollection 2020. PMID 32582758
- [Derived] Staehler M, Motzer RJ, George DJ, Pandha HS, Donskov F, Escudier B, Pantuck AJ, Patel A, DeAnnuntis L, Bhattacharyya H, Ramaswamy K, Zanotti G, Lin X, Lechuga M, Serfass L, Paty J, Ravaud A. Adjuvant sunitinib in patients with high-risk renal cell carcinoma: safety, therapy management, and patient-reported outcomes in the S-TRAC trial. Ann Oncol. 2018 Oct 1;29(10):2098-2104. doi: 10.1093/annonc/mdy329. PMID 30412222
- [Derived] Rini BI, Escudier B, Martini JF, Magheli A, Svedman C, Lopatin M, Knezevic D, Goddard AD, Febbo PG, Li R, Lin X, Valota O, Staehler M, Motzer RJ, Ravaud A. Validation of the 16-Gene Recurrence Score in Patients with Locoregional, High-Risk Renal Cell Carcinoma from a Phase III Trial of Adjuvant Sunitinib. Clin Cancer Res. 2018 Sep 15;24(18):4407-4415. doi: 10.1158/1078-0432.CCR-18-0323. Epub 2018 May 17. PMID 29773662
- [Derived] George DJ, Martini JF, Staehler M, Motzer RJ, Magheli A, Escudier B, Gerletti P, Li S, Casey M, Laguerre B, Pandha HS, Pantuck AJ, Patel A, Lechuga MJ, Ravaud A. Immune Biomarkers Predictive for Disease-Free Survival with Adjuvant Sunitinib in High-Risk Locoregional Renal Cell Carcinoma: From Randomized Phase III S-TRAC Study. Clin Cancer Res. 2018 Apr 1;24(7):1554-1561. doi: 10.1158/1078-0432.CCR-17-2822. Epub 2018 Jan 26. PMID 29374054
- [Derived] Motzer RJ, Ravaud A, Patard JJ, Pandha HS, George DJ, Patel A, Chang YH, Escudier B, Donskov F, Magheli A, Carteni G, Laguerre B, Tomczak P, Breza J, Gerletti P, Lechuga M, Lin X, Casey M, Serfass L, Pantuck AJ, Staehler M. Adjuvant Sunitinib for High-risk Renal Cell Carcinoma After Nephrectomy: Subgroup Analyses and Updated Overall Survival Results. Eur Urol. 2018 Jan;73(1):62-68. doi: 10.1016/j.eururo.2017.09.008. Epub 2017 Sep 28. PMID 28967554
- [Derived] Ravaud A, Motzer RJ, Pandha HS, George DJ, Pantuck AJ, Patel A, Chang YH, Escudier B, Donskov F, Magheli A, Carteni G, Laguerre B, Tomczak P, Breza J, Gerletti P, Lechuga M, Lin X, Martini JF, Ramaswamy K, Casey M, Staehler M, Patard JJ; S-TRAC Investigators. Adjuvant Sunitinib in High-Risk Renal-Cell Carcinoma after Nephrectomy. N Engl J Med. 2016 Dec 8;375(23):2246-2254. doi: 10.1056/NEJMoa1611406. Epub 2016 Oct 9. PMID 27718781

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 674 enrolled participants (615 in global cohort and 59 in china cohort), the results presented refers to the study conducted on 615 (intent-to-treat population) in 21 countries and were randomized to sunitinib and placebo for 9 cycles (1 cycle=42 days).
Pre-assignment Details: Screening: From Week 0 (nephrectomy surgery) to Week 11; in this period, echocardiogram/multi-gated acquisition, post-surgery imaging, histopathology, physical examination, laboratory tests, electrocardiogram and concomitant treatment were assessed. Randomization occurred not before 3 weeks post-nephrectomy & not after 12 weeks post-nephrectomy.
Groups:
- Sunitinib: Participants received Sunitinib on 9 6-week cycles on 4/2 dosing schedule: 4 weeks on, 2 weeks off.
- Placebo: Participants received Placebo on 9 6-week cycles with 4/2 dosing schedule: 4 weeks on, 2 weeks off.
Period: Overall Study
Arm/Group | Sunitinib | Placebo
Started | 309 | 306
Intent-to-Treat Population (All randomized participants, who received study drug/a different drug to which they were randomized) | 309 | 306
As-Treated Population (All participants, who received at least 1 dose of study drug according to actual study treatment) | 306 (3 were randomized but not treated: 2 refused treatment & 1 withdrew before receiving study drug) | 304 (2 were randomized but not treated: 1 was screening failure & 1 discontinued due to new liver lesions)
Completed | 165 | 165
Not Completed | 144 | 141
Not completed — Other | 26 | 18
Not completed — Death | 67 | 76
Not completed — Participants refused further follow-up | 31 | 30
Not completed — Lost to Follow-up | 17 | 15
Not completed — Enrolled but not treated | 3 | 2

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population included all participants who were randomized, with study drug assignment designated according to initial randomization, regardless of whether participants received study drug or received a different drug from that to which they were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sunitinib | Placebo | Total
Number analyzed (Participants) | 309 | 306 | 615
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (10.6) | 57.9 (10.6) | 57.9 (10.6)
Age, Customized [Number; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 233 | 224 | 457
  >=65 years | 76 | 82 | 158
Sex/Gender, Customized [Number; unit: Participants]
  Female | 87 | 77 | 164
  Male | 222 | 229 | 451

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival (DFS)- Assessed by Blinded Independent Central Review
Description: DFS was defined as the time interval (in years) from the date of randomization to the first date of recurrence or occurrence of a secondary malignancy or death. Recurrence refers to relapse of the primary tumor in-situ or at metastatic sites. Date of recurrence or occurrence: The date of the recurrence or occurrence of a secondary malignancy for the first time, either by blinded independent central review (BICR) or investigator assessment for respective analyses. Participants were followed with tumor imaging for recurrence or occurrence of a secondary malignancy for remainder of follow-up period unless the participant had withdrawn consent. According to the statistical analysis plan there are two cohorts: 1.Global Cohort: primary analysis of DFS was performed approximately 5 years after last participant in the Global Cohort is randomized; 2. China Cohort: primary analysis of DFS was performed approximately 3 years after the last participant in China Cohort was randomized.
Time Frame: Every 12 weeks during the first 3 years and every 6 months after that unless the participant had withdrawn consent. Performed 5 years after LSLV or when approximately 258 events survival status, whichever was later.
Population: ITT population included all participants who were randomized, with study drug assignment designated according to initial randomization, regardless of whether participants received study drug or received a different drug from that to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Number of years
Arm/Group | Sunitinib | Placebo
Number analyzed (Participants) | 309 | 306
Number of years | 6.8 [5.8 to NA] — The upper limit of the 95% confidence interval of the median DFS on Sunitinib was not reached | 5.6 [3.8 to 6.6]
Statistical Analysis 1: Comparison: Sunitinib vs Placebo; Superiority analysis; Test type: Superiority; p = 0.030, Cox Proportional hazards model; Based on the Cox Proportional hazards model stratified by UISS High-Risk Group; Cox Proportional Hazard = 0.761, 95% CI 2-sided [0.594 to 0.975]

2. Primary Outcome: DFS- Assessed by the Investigator [Stratified by University of California Los Angeles Integrated Staging System (UISS) High Risk Group-Intent to Treat Population]
Description: DFS was defined as the time interval (in years) from the date of randomization to the first date of recurrence or occurrence of a secondary malignancy or death. Recurrence refers to relapse of the primary tumor in-situ or at metastatic sites.
  Date of recurrence or occurrence: The date of the recurrence or occurrence of a secondary malignancy for the first time, either by BICR or investigator assessment for the respective analyses.
  Participants were followed with tumor imaging for recurrence or occurrence of a secondary malignancy for the remainder of the follow-up period unless the participants had withdrawn consent.
  According to the statistical analysis plan there are two cohorts: 1.Global Cohort: primary analysis of DFS was performed approximately 5 years after last participant in the Global Cohort is randomized; 2. China Cohort: primary analysis of DFS was performed approximately 3 years after the last participant in China Cohort was randomized.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Number of years
Arm/Group | Sunitinib | Placebo
Number analyzed (Participants) | 309 | 306
Number of years | 6.5 [4.7 to 7.0] | 4.5 [3.8 to 5.9]
Statistical Analysis 1: Comparison: Sunitinib vs Placebo; Superiority analysis; Test type: Superiority; p = 0.077, Cox Proportional hazards model; Based on the Cox Proportional hazards model stratified by UISS High-Risk Group; Cox Proportional Hazard = 0.811, 95% CI 2-sided [0.643 to 1.023]

3. Secondary Outcome: Overall Survival (OS)- (Stratified by UISS High Risk Group-Intent to Treat Population)
Description: OS was defined as the time from the date of randomization to the date of death due to any cause.
Time Frame: Every 12 weeks until the time for final analysis (up to data cut-off date: 30 April 2017; maximum exposure:14.9 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Year
Arm/Group | Sunitinib | Placebo
Number analyzed (Participants) | 309 | 306
Year | NA [NA to NA] — Data was not estimable due to small number of participants with an event. | NA [NA to NA] — Data was not estimable due to small number of participants with an event.
Statistical Analysis 1: Comparison: Sunitinib vs Placebo; Hazard ratio was based on the Cox Proportional hazards model stratified by UISS High-Risk Group; Test type: Superiority; p = 0.661, Log-rank test; Hazard Ratio (HR) = 0.929, 95% CI 2-sided [0.670 to 1.289]

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) by Severity
Description: TEAEs are all AEs (serious and non-serious) occurred, for the first time, on or after the first day of study treatment. AEs started before the first dose of study treatment but increased in severity (CTC grade) over the baseline will also be considered TEAEs.
  Participants were followed for AEs from the first day of study treatment until at least 28 days after the last on-study treatment administration, or until all serious or study medication-related toxicities had resolved or were determined to be "chronic" or "stable," whichever was later. The treatment was administered to the participants from cycle1/day 1 up to 9 cycles or until relapse, secondary malignancy, death or withdraw for other reasons such as toxicity or withdraw of consent.
Time Frame: Cycle 1(Day 1 & Day 28); subsequent cycles (Day 1); end of treatment/withdrawal and 28 days post treatment, or until all serious or study medication-related toxicities had resolved or were determined to be "chronic" or "stable," whichever was later
Population: The As-Treated (AT) population included all participants who received at least 1 dose of study drug with treatment assignments designated according to actual study treatment received. This population was the primary population for evaluating treatment administration/ compliance and safety.
Measure: Number; unit: Number of participants
Arm/Group | Sunitinib | Placebo
Number analyzed (Participants) | 306 | 304
Number of participants
  Participants With Adverse Events (AEs) | 305 | 270
  Participants With Serious Adverse Events (SAEs) | 67 | 52
  Participants With Grade 3 or 4 AEs | 189 | 61
  Participants With Grade 5 AEs | 5 | 5
  Participants Discontinued Due to AEs | 86 | 16
  Participants With Dose Reduced Due to AEs | 106 | 6
  Temporary Discontinuation Due to AEs | 141 | 40

5. Secondary Outcome: Summary of Duration of Treatment-Emergent Adverse Events of Special Interest by MedDRA Preferred Terms (All Causalities, All Cycles)
Description: as for outcome 4
Time Frame: as for outcome 4
Population: AT population: All participants who received at least 1 dose of study drug with treatment assignments designated according to actual study treatment received.
  The numbers of participants analyzed were the participants with any adverse event of special interest (AESI) and that one participant could have reported more than one AESI
Measure: Mean (Standard Deviation); unit: Weeks
Arm/Group | Sunitinib | Placebo
Number analyzed (Participants) | 306 | 304
Weeks
  Benign Neoplasm of Thyroid Gland: number analyzed (Participants) | 0 | 1
  Benign Neoplasm of Thyroid Gland |  | 35.1
  Goitre: number analyzed (Participants) | 0 | 2
  Goitre |  | 305.6 (97.08)
  Hyperthyroidism: number analyzed (Participants) | 12 | 2
  Hyperthyroidism | 23.2 (25.95) | 110.8 (146.57)
  Hypothyroidism: number analyzed (Participants) | 56 | 4
  Hypothyroidism | 46.9 (75.30) | 58.0 (62.06)
  Papillary Thyroid Cancer: number analyzed (Participants) | 0 | 1
  Papillary Thyroid Cancer |  | 22.1
  Thyroid Disorder: number analyzed (Participants) | 1 | 0
  Thyroid Disorder | 19 |
  Thyroid Mass: number analyzed (Participants) | 0 | 1
  Thyroid Mass |  | 20.4

6. Secondary Outcome: Patient-Reported Outcomes (PROs)- European Organization for Research and Treatment of Cancer (EORTC) QLQ C30: Observed Means in Global Health Status / Quality of Life Scale Scores
Description: Patient-reported outcomes (PROs) assessed health-related quality of life (QoL) by using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30), which was a 30-item questionnaire with global QoL scale, 5 multi-item functional scales (physical, role, emotional, cognitive, & social functioning), 3 multi-item symptom scales (fatigue, nausea/vomiting, & pain), and 6 single item symptom scales for other cancer-related symptoms (dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, & the financial impact of cancer). The questionnaire includes 28 items with 4-point Likert type responses from "not at all" to "very much" to assess functioning & symptoms; 2 items with 7-point Likert scales for global health & overall QoL. All responses were converted to a 0 to 100 scale using a standard scoring algorithm, higher scores represented better level for functioning/QoL & more severe for symptoms.
Time Frame: Cycle 1(Day 1); subsequent cycles (Day 1) and end of treatment/withdrawal (ie, up to 1 year)
Population: ITT population included all participants who were randomized, with study drug assignment designated according to initial randomization, regardless of whether participants received study drug or a different drug from that to which they were randomized. Here, 'Number analyzed' signifies the number of participants evaluable at specified time-points.
Measure: Mean (Standard Error); unit: Scores on scale
Arm/Group | Sunitinib | Placebo
Number analyzed (Participants) | 309 | 306
Scores on scale
  Cycle 1 (Baseline): number analyzed (Participants) | 292 | 288
  Cycle 1 (Baseline) | 74.83 (1.044) | 75.61 (1.044)
  Cycle 2: number analyzed (Participants) | 260 | 274
  Cycle 2 | 69.71 (1.289) | 75.49 (1.097)
  Cycle 3: number analyzed (Participants) | 241 | 265
  Cycle 3 | 69.67 (1.278) | 74.09 (1.142)
  Cycle 4: number analyzed (Participants) | 227 | 249
  Cycle 4 | 66.52 (1.307) | 74.93 (1.109)
  Cycle 5: number analyzed (Participants) | 219 | 234
  Cycle 5 | 68.34 (1.340) | 74.61 (1.179)
  Cycle 6: number analyzed (Participants) | 210 | 231
  Cycle 6 | 66.27 (1.396) | 75.69 (1.172)
  Cycle 7: number analyzed (Participants) | 200 | 220
  Cycle 7 | 67.42 (1.447) | 73.98 (1.222)
  Cycle 8: number analyzed (Participants) | 185 | 212
  Cycle 8 | 68.33 (1.376) | 74.49 (1.260)
  Cycle 9: number analyzed (Participants) | 177 | 203
  Cycle 9 | 68.31 (1.556) | 74.06 (1.338)
  End of treatment (EOT): number analyzed (Participants) | 250 | 250
  End of treatment (EOT) | 64.43 (1.367) | 73.37 (1.264)

7. Secondary Outcome: PROs- EORTC QLQ C30: Functional Scale Scores Between Treatment Comparison
Description: Patient-reported outcomes (PROs) assessed health-related quality of life (QoL) by using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30), which was a 30-item questionnaire with global QoL scale & 5 multi-item functional scales (physical, role, emotional, cognitive, & social functioning). The questionnaire includes 28 items with 4-point Likert type responses from "not at all" to "very much" to assess functioning; 2 items with 7-point Likert scales for global health & overall QoL. All responses were converted to a 0 to 100 scale using a standard scoring algorithm, higher scores represented better level for functioning/QoL.
Time Frame: Cycle 1(Day 1); subsequent cycles (Day 1) and end of treatment/withdrawal (ie, up to 1 year)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Scores on scale
Arm/Group | Sunitinib | Placebo
Number analyzed (Participants) | 309 | 306
Scores on scale
  Physical | 83.54 [82.40 to 84.68] | 87.53 [86.42 to 88.64]
  Role | 78.94 [77.14 to 80.74] | 85.46 [83.70 to 87.23]
  Emotional | 80.92 [79.58 to 82.27] | 82.97 [81.66 to 84.29]
  Cognitive | 85.50 [84.17 to 86.83] | 87.43 [86.13 to 88.73]
  Social | 80.62 [79.04 to 82.21] | 87.99 [86.44 to 89.53]

8. Secondary Outcome: PROs- EORTC QLQ-C30: Symptom Scale Scores Between Treatment Comparison
Description: PROs assessed health-related QoL by using the EORTC QLQ-C30, which was a 30 multi-item symptom scales (fatigue, nausea/vomiting, & pain), and 6 single item symptom scales for other cancer-related symptoms (dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, & the financial impact of cancer). The questionnaire includes 28 items with 4-point Likert type responses from "not at all" to "very much" to assess symptoms. All responses were converted to a 0 to 100 scale using a standard scoring algorithm, higher scores represented more severe symptoms.
Time Frame: Cycle 1(Day 1); subsequent cycles (Day 1) and end of treatment/withdrawal (ie, up to 1 year)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Scores on scale
Arm/Group | Sunitinib | Placebo
Number analyzed (Participants) | 309 | 306
Scores on scale
  Fatigue | 29.94 [28.33 to 31.56] | 21.74 [20.16 to 23.31]
  Nausea and Vomiting | 7.35 [6.38 to 8.33] | 3.46 [2.51 to 4.41]
  Pain | 21.81 [20.10 to 23.52] | 16.63 [14.96 to 18.30]
  Dyspnoea | 14.97 [13.38 to 16.57] | 11.89 [10.33 to 13.45]
  Insomnia | 22.22 [20.26 to 24.19] | 20.73 [18.81 to 22.65]
  Appetite Loss | 14.66 [13.12 to 16.21] | 4.62 [3.11 to 6.13]
  Constipation | 11.24 [9.66 to 12.82] | 9.83 [8.29 to 11.37]
  Diarrhoea | 19.25 [17.54 to 20.95] | 7.25 [5.59 to 8.91]
  Financial Difficulties | 15.12 [13.42 to 16.82] | 13.92 [12.26 to 15.59]

9. Secondary Outcome: PROs- EuroQoL EQ-5D Observed Means - Intent to Treat Population
Description: Patient-reported outcomes (PROs) assessed health-related quality of life (QoL) by the EuroQoL Group health status questionnaire (EQ-5D), which was a brief self-administered, validated instrument with 2 parts. In this outcome measure, the first part with 5 descriptors of current health state (mobility, self-care, usual activities, pain/discomfort, & anxiety/depression) was used; a participant was asked to rate each state on a 3-level scale (1=no problem, 2=some problem, & 3=extreme problem); higher levels indicated greater severity/impairment. The published weights allowed the creation of a single summary score called the EQ-5D index, which ranged from -0.594 to 1; low scores represented a higher level of dysfunction & 1 as perfect health.
Time Frame: Cycle 1(Day 1); subsequent cycles (Day 1) and end of treatment/withdrawal (ie, up to 1 year)
Population: as for outcome 6
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Sunitinib | Placebo
Number analyzed (Participants) | 309 | 306
Units on a scale
  Cycle 1 (Baseline): number analyzed (Participants) | 293 | 287
  Cycle 1 (Baseline) | 0.84 (0.011) | 0.83 (0.011)
  Cycle 2: number analyzed (Participants) | 255 | 271
  Cycle 2 | 0.83 (0.011) | 0.84 (0.011)
  Cycle 3: number analyzed (Participants) | 235 | 267
  Cycle 3 | 0.80 (0.013) | 0.82 (0.012)
  Cycle 4: number analyzed (Participants) | 231 | 245
  Cycle 4 | 0.77 (0.014) | 0.84 (0.011)
  Cycle 5: number analyzed (Participants) | 218 | 230
  Cycle 5 | 0.77 (0.016) | 0.84 (0.013)
  Cycle 6: number analyzed (Participants) | 211 | 234
  Cycle 6 | 0.78 (0.016) | 0.85 (0.012)
  Cycle 7: number analyzed (Participants) | 199 | 216
  Cycle 7 | 0.77 (0.016) | 0.83 (0.014)
  Cycle 8: number analyzed (Participants) | 185 | 207
  Cycle 8 | 0.80 (0.015) | 0.84 (0.013)
  Cycle 9: number analyzed (Participants) | 174 | 202
  Cycle 9 | 0.81 (0.015) | 0.85 (0.013)
  EOT: number analyzed (Participants) | 250 | 245
  EOT | 0.75 (0.017) | 0.83 (0.015)

10. Secondary Outcome: PROs- EuroQol European Quality of Life Questionnaire Variable Analogue Scale (EQ-VAS) Observed Means
Description: Patient-reported outcomes (PROs) assessed health-related quality of life (QoL) by the EuroQoL Group health status questionnaire (EQ-5D), which was a brief self-administered, validated instrument with 2 parts. The first part assessed the current health state. In this outcome measure, the second part was applied to assess the general health status by using visual analog scale (EQ-5D VAS) which measured participant's self-rated health status on a scale ranging from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: Cycle 1(Day 1); subsequent cycles (Day 1) and end of treatment/withdrawal (ie, up to 1 year)
Population: as for outcome 6
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Sunitinib | Placebo
Number analyzed (Participants) | 309 | 306
Units on a scale
  Cycle 1 (Baseline): number analyzed (Participants) | 293 | 287
  Cycle 1 (Baseline) | 77.31 (0.999) | 75.67 (1.080)
  Cycle 2: number analyzed (Participants) | 261 | 268
  Cycle 2 | 74.39 (1.188) | 76.99 (1.080)
  Cycle 3: number analyzed (Participants) | 234 | 261
  Cycle 3 | 74.20 (1.093) | 76.85 (1.122)
  Cycle 4: number analyzed (Participants) | 231 | 246
  Cycle 4 | 74.14 (1.118) | 77.34 (1.115)
  Cycle 5: number analyzed (Participants) | 218 | 233
  Cycle 5 | 73.30 (1.220) | 77.56 (1.212)
  Cycle 6: number analyzed (Participants) | 211 | 232
  Cycle 6 | 73.51 (1.250) | 78.61 (1.130)
  Cycle 7: number analyzed (Participants) | 199 | 218
  Cycle 7 | 72.27 (1.267) | 77.49 (1.180)
  Cycle 8: number analyzed (Participants) | 186 | 209
  Cycle 8 | 73.96 (1.226) | 77.65 (1.213)
  Cycle 9: number analyzed (Participants) | 174 | 203
  Cycle 9 | 72.93 (1.424) | 79.02 (1.168)
  EOT: number analyzed (Participants) | 251 | 246
  EOT | 71.79 (1.139) | 76.93 (1.283)

11. Secondary Outcome: Number of Participants With Tolerability Symptoms
Description: Participants were followed for AEs from the first day of study treatment until at least 28 days after the last on-study treatment administration, or until all serious or study medication-related toxicities had resolved or were determined to be "chronic" or "stable," whichever was later.
  The treatment was administered to the participants from cycle1/day 1 up to 9 cycles or until relapse, secondary malignancy, death or withdraw for other reasons such as toxicity or withdraw of consent. This table provides the summary of discontinuations de to adverse events. Participants were counted only once in each row.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Number; unit: Number of participants
Arm/Group | Sunitinib | Placebo
Number analyzed (Participants) | 309 | 306
Number of participants
  Palmar-plantar erythrodysaesthesia syndrome | 13 | 0
  Hypertension | 6 | 0
  Asthenia | 4 | 0
  Fatigue | 3 | 1
  Pulmonary embolism | 3 | 1
  Gastrooesophageal reflux disease | 3 | 0
  Ejection fraction decreased | 2 | 1
  Left ventricular dysfunction | 2 | 1
  Acute myocardial infarction | 2 | 0
  Blood creatinine increased | 2 | 0
  Dehydration | 2 | 0
  Dyspepsia | 2 | 0
  Proteinuria | 2 | 0
  Thrombocytopenia | 2 | 0
  Upper gastrointestinal haemorrhage | 2 | 0
  Vomiting | 2 | 0
  Electrocardiogram QT prolonged | 1 | 1
  Lethargy | 1 | 1
  Transient ischaemic attack | 1 | 1
  Depression | 0 | 2
  Abdominal pain | 1 | 0
  Abdominal pain upper | 1 | 0
  Acute kidney injury | 1 | 0
  Ageusia | 1 | 0
  Alanine aminotransferase increased | 1 | 0
  Anal inflammation | 1 | 0
  Anal pruritus | 1 | 0
  Aspartate aminotransferase increased | 1 | 0
  Atrial fibrillation | 1 | 0
  Atrial flutter | 1 | 0
  Diarrhoea | 1 | 0
  Disease progression | 1 | 0
  Dysgeusia | 1 | 0
  Electrocardiogram ST segment abnormal | 1 | 0
  Embolism venous | 1 | 0
  Eyelid oedema | 1 | 0
  Gastritis haemorrhagic | 1 | 0
  Glossodynia | 1 | 0
  Hepatic function abnormal | 1 | 0
  Hepatitis acute | 1 | 0
  Hypercreatininaemia | 1 | 0
  Hypertransaminasaemia | 1 | 0
  Hypothyroidism | 1 | 0
  Influenza like illness | 1 | 0
  Mental status changes | 1 | 0
  Mucosal inflammation | 1 | 0
  Myalgia | 1 | 0
  Myocardial infarction | 1 | 0
  Myocarditis | 1 | 0
  Necrosis | 1 | 0
  Nephrotic syndrome | 1 | 0
  Neutropenia | 1 | 0
  Oedema peripheral | 1 | 0
  Pancytopenia | 1 | 0
  Post procedural infection | 1 | 0
  Presyncope | 1 | 0
  Pyrexia | 1 | 0
  Stomatitis | 1 | 0
  Therapeutic response unexpected | 1 | 0
  Tremor | 1 | 0
  Vena cava thrombosis | 1 | 0
  Vertigo | 1 | 0
  Agitated depression | 0 | 1
  Angina unstable | 0 | 1
  Brain cancer metastatic | 0 | 1
  Hepatitis | 0 | 1
  Hypersensitivity | 0 | 1
  Metastases to lung | 0 | 1
  Mood altered | 0 | 1
  Renal impairment | 0 | 1
  Tinnitus | 0 | 1

ADVERSE EVENTS:
Time Frame: Cycle 1(Day 1 & Day 28); subsequent cycles (Day 1); end of treatment/withdrawal and 28 days post-treatment, or until all serious or study medication-related toxicities had resolved or were determined to be "chronic" or "stable," whichever was later.
Description: Participants were followed for AEs from the first day of study treatment until at least 28 days after the last on-study treatment administration, or until all serious or study medication-related toxicities had resolved or were determined to be "chronic" or "stable," whichever was later.
Arm/Group | Sunitinib | Placebo
All-Cause Mortality (participants affected / at risk) | 67/306 | 76/304
Serious Adverse Events (participants affected / at risk) | 67/306 | 52/304
Other Adverse Events (participants affected / at risk) | 303/306 | 270/304
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=306) | Placebo (N=304)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 2 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 3 | 1
Myocarditis (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 2 | 1
Disease progression (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 2 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Pyrexia (General disorders) | 5 | 0
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 2 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Bronchitis viral (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Pneumonia legionella (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 3
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carcinoid tumour of the gastrointestinal tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Axonal neuropathy (Nervous system disorders) | 1 | 0
Cerebral haematoma (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Headache (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 1
Agitated depression (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 2
Mental status changes (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Albuminuria (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 1
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Gastrectomy (Surgical and medical procedures) | 0 | 1
Splenectomy (Surgical and medical procedures) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 8 | 2
Orthostatic hypotension (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Vena cava thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=306) | Placebo (N=304)
Anaemia (Blood and lymphatic system disorders) | 33 | 7
Eosinopenia (Blood and lymphatic system disorders) | 1 | 0
Hyperglobulinaemia (Blood and lymphatic system disorders) | 0 | 1
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 45 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 8 | 1
Monocytopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 70 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 61 | 4
Angina pectoris (Cardiac disorders) | 5 | 1
Aortic valve stenosis (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 2 | 5
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 5
Bradycardia (Cardiac disorders) | 1 | 1
Bundle branch block left (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 2
Cardiovascular disorder (Cardiac disorders) | 0 | 1
Conduction disorder (Cardiac disorders) | 1 | 0
Diastolic dysfunction (Cardiac disorders) | 1 | 0
Extrasystoles (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 7 | 3
Left ventricular hypertrophy (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 1
Mitral valve prolapse (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 3
Pericardial effusion (Cardiac disorders) | 2 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 2 | 2
Supraventricular extrasystoles (Cardiac disorders) | 1 | 2
Tachycardia (Cardiac disorders) | 1 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 1
Ventricular hypokinesia (Cardiac disorders) | 1 | 0
Dermoid cyst (Congenital, familial and genetic disorders) | 0 | 1
Deafness (Ear and labyrinth disorders) | 1 | 1
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 3 | 1
External ear pain (Ear and labyrinth disorders) | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 3 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 5 | 5
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 8 | 12
Goitre (Endocrine disorders) | 0 | 2
Hyperparathyroidism (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 12 | 2
Hypothyroidism (Endocrine disorders) | 56 | 4
Oestrogen deficiency (Endocrine disorders) | 0 | 1
Thyroid disorder (Endocrine disorders) | 1 | 0
Thyroid mass (Endocrine disorders) | 0 | 1
Blindness unilateral (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 3 | 1
Cataract subcapsular (Eye disorders) | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 2 | 0
Diplopia (Eye disorders) | 2 | 0
Dry eye (Eye disorders) | 4 | 1
Eye discharge (Eye disorders) | 1 | 0
Eye haemorrhage (Eye disorders) | 2 | 0
Eye inflammation (Eye disorders) | 0 | 1
Eye irritation (Eye disorders) | 5 | 0
Eye oedema (Eye disorders) | 7 | 0
Eye pain (Eye disorders) | 3 | 0
Eye pruritus (Eye disorders) | 1 | 1
Eye swelling (Eye disorders) | 2 | 0
Eyelash discolouration (Eye disorders) | 2 | 0
Eyelid bleeding (Eye disorders) | 1 | 0
Eyelid oedema (Eye disorders) | 21 | 1
Eyelid pain (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 1 | 1
Lacrimal disorder (Eye disorders) | 0 | 1
Lacrimal gland enlargement (Eye disorders) | 0 | 1
Lacrimation increased (Eye disorders) | 12 | 1
Ocular hyperaemia (Eye disorders) | 1 | 0
Ocular surface disease (Eye disorders) | 1 | 0
Oscillopsia (Eye disorders) | 1 | 0
Periorbital oedema (Eye disorders) | 7 | 0
Photophobia (Eye disorders) | 2 | 0
Photopsia (Eye disorders) | 0 | 1
Retinopathy hypertensive (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 2 | 3
Visual acuity reduced (Eye disorders) | 1 | 1
Visual impairment (Eye disorders) | 4 | 1
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 8 | 8
Abdominal distension (Gastrointestinal disorders) | 11 | 4
Abdominal hernia (Gastrointestinal disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 42 | 15
Abdominal pain lower (Gastrointestinal disorders) | 7 | 1
Abdominal pain upper (Gastrointestinal disorders) | 40 | 13
Abdominal rigidity (Gastrointestinal disorders) | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0
Abnormal faeces (Gastrointestinal disorders) | 2 | 0
Anal fissure (Gastrointestinal disorders) | 2 | 0
Anal haemorrhage (Gastrointestinal disorders) | 2 | 0
Anal inflammation (Gastrointestinal disorders) | 6 | 0
Anal pruritus (Gastrointestinal disorders) | 3 | 0
Anal skin tags (Gastrointestinal disorders) | 1 | 0
Anorectal discomfort (Gastrointestinal disorders) | 4 | 1
Anorectal disorder (Gastrointestinal disorders) | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 12 | 2
Bowel movement irregularity (Gastrointestinal disorders) | 1 | 0
Breath odour (Gastrointestinal disorders) | 0 | 2
Change of bowel habit (Gastrointestinal disorders) | 1 | 0
Chapped lips (Gastrointestinal disorders) | 2 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 36 | 32
Dental caries (Gastrointestinal disorders) | 4 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 14 | 8
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 1
Duodenogastric reflux (Gastrointestinal disorders) | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 82 | 19
Dysphagia (Gastrointestinal disorders) | 15 | 1
Eructation (Gastrointestinal disorders) | 4 | 1
Flatulence (Gastrointestinal disorders) | 26 | 14
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 | 1
Gastric mucosa erythema (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 5 | 4
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 2
Gastrointestinal dysplasia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal hypermotility (Gastrointestinal disorders) | 2 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 27 | 9
Gingival bleeding (Gastrointestinal disorders) | 9 | 0
Gingival oedema (Gastrointestinal disorders) | 1 | 0
Gingival pain (Gastrointestinal disorders) | 2 | 1
Gingival recession (Gastrointestinal disorders) | 1 | 0
Gingival swelling (Gastrointestinal disorders) | 2 | 0
Gingival ulceration (Gastrointestinal disorders) | 1 | 0
Glossitis (Gastrointestinal disorders) | 4 | 1
Glossodynia (Gastrointestinal disorders) | 4 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 12 | 3
Hiatus hernia (Gastrointestinal disorders) | 1 | 1
Hyperchlorhydria (Gastrointestinal disorders) | 3 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 4 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Lip disorder (Gastrointestinal disorders) | 1 | 0
Lip dry (Gastrointestinal disorders) | 0 | 1
Lip ulceration (Gastrointestinal disorders) | 1 | 0
Loose tooth (Gastrointestinal disorders) | 1 | 0
Mouth cyst (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 9 | 3
Nausea (Gastrointestinal disorders) | 103 | 42
Odynophagia (Gastrointestinal disorders) | 5 | 0
Oesophageal pain (Gastrointestinal disorders) | 3 | 0
Oesophagitis (Gastrointestinal disorders) | 14 | 1
Oral discomfort (Gastrointestinal disorders) | 4 | 0
Oral disorder (Gastrointestinal disorders) | 3 | 0
Oral mucosal blistering (Gastrointestinal disorders) | 1 | 0
Oral mucosal erythema (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 7 | 2
Oral toxicity (Gastrointestinal disorders) | 1 | 0
Palatal oedema (Gastrointestinal disorders) | 1 | 0
Palatal swelling (Gastrointestinal disorders) | 0 | 1
Pancreatic steatosis (Gastrointestinal disorders) | 0 | 1
Perianal erythema (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 7 | 1
Proctitis (Gastrointestinal disorders) | 9 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 6 | 1
Regurgitation (Gastrointestinal disorders) | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 2 | 0
Sensitivity of teeth (Gastrointestinal disorders) | 2 | 1
Stomatitis (Gastrointestinal disorders) | 81 | 13
Swollen tongue (Gastrointestinal disorders) | 1 | 1
Tongue disorder (Gastrointestinal disorders) | 1 | 0
Tongue oedema (Gastrointestinal disorders) | 1 | 0
Tongue ulceration (Gastrointestinal disorders) | 3 | 1
Tooth loss (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 5 | 3
Vomiting (Gastrointestinal disorders) | 55 | 20
Asthenia (General disorders) | 69 | 36
Chest discomfort (General disorders) | 4 | 2
Chest pain (General disorders) | 11 | 13
Chills (General disorders) | 10 | 4
Cyst (General disorders) | 1 | 0
Death (General disorders) | 1 | 0
Face oedema (General disorders) | 28 | 1
Facial pain (General disorders) | 1 | 0
Fatigue (General disorders) | 112 | 74
Feeling abnormal (General disorders) | 1 | 0
Feeling cold (General disorders) | 4 | 2
Feeling hot (General disorders) | 0 | 2
Feeling of body temperature change (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 3 | 2
Generalised oedema (General disorders) | 1 | 0
Hernia (General disorders) | 1 | 2
Hypothermia (General disorders) | 1 | 1
Impaired healing (General disorders) | 1 | 0
Influenza like illness (General disorders) | 11 | 5
Infusion site extravasation (General disorders) | 0 | 1
Injection site haematoma (General disorders) | 1 | 0
Injection site inflammation (General disorders) | 0 | 1
Localised oedema (General disorders) | 2 | 0
Malaise (General disorders) | 6 | 1
Mucosal discolouration (General disorders) | 0 | 1
Mucosal dryness (General disorders) | 4 | 1
Mucosal induration (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 102 | 25
Necrosis (General disorders) | 1 | 0
Oedema (General disorders) | 10 | 2
Oedema mucosal (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 24 | 16
Pain (General disorders) | 9 | 9
Peripheral swelling (General disorders) | 3 | 0
Pyrexia (General disorders) | 32 | 17
Secretion discharge (General disorders) | 1 | 0
Swelling (General disorders) | 1 | 0
Temperature intolerance (General disorders) | 4 | 0
Therapeutic response unexpected (General disorders) | 1 | 0
Xerosis (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 5 | 2
Hypertransaminasaemia (Hepatobiliary disorders) | 2 | 1
Jaundice (Hepatobiliary disorders) | 20 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Contrast media allergy (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 3 | 5
Seasonal allergy (Immune system disorders) | 1 | 0
Angular cheilitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 6 | 6
Bronchitis viral (Infections and infestations) | 1 | 0
Candida infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 3 | 0
Conjunctivitis (Infections and infestations) | 8 | 4
Cystitis (Infections and infestations) | 3 | 2
Diverticulitis (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 2 | 4
Enteritis infectious (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 1
Eye infection (Infections and infestations) | 0 | 2
Folliculitis (Infections and infestations) | 0 | 1
Fungal infection (Infections and infestations) | 3 | 0
Fungal skin infection (Infections and infestations) | 1 | 2
Gastroenteritis (Infections and infestations) | 2 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 2
Genital candidiasis (Infections and infestations) | 1 | 0
Genital herpes (Infections and infestations) | 1 | 0
Gingivitis (Infections and infestations) | 8 | 0
Helicobacter gastritis (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0
Herpes virus infection (Infections and infestations) | 5 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Hordeolum (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 6 | 3
Liver abscess (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 3 | 0
Laryngitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 4
Lung infection (Infections and infestations) | 1 | 1
Oral herpes (Infections and infestations) | 7 | 3
Oral infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 15 | 20
Osteomyelitis (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 2 | 0
Periodontitis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 6 | 5
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Pilonidal cyst (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Post procedural infection (Injury, poisoning and procedural complications) | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1
Pulpitis dental (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 2
Retinitis (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 7 | 3
Rhinolaryngitis (Infections and infestations) | 1 | 0
Sinobronchitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 4 | 2
Skin infection (Infections and infestations) | 2 | 0
Staphylococcal scalded skin syndrome (Infections and infestations) | 1 | 0
Tinea pedis (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 2 | 0
Tooth infection (Infections and infestations) | 3 | 2
Tracheitis (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 6 | 5
Urinary tract infection (Infections and infestations) | 7 | 7
Urogenital infection fungal (Infections and infestations) | 1 | 0
Vaginal infection (Infections and infestations) | 2 | 1
Viral hepatitis carrier (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 4 | 0
Viral labyrinthitis (Infections and infestations) | 0 | 1
Vulvitis (Infections and infestations) | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 1
Wound infection (Infections and infestations) | 0 | 1
Burn oesophageal (Injury, poisoning and procedural complications) | 1 | 1
Burn oral cavity (Injury, poisoning and procedural complications) | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 7 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 2
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 7
Laceration (Injury, poisoning and procedural complications) | 1 | 3
Ligament injury (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 2
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Infections and infestations) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 2 | 5
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Skin injury (Injury, poisoning and procedural complications) | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0
Stress fracture (Injury, poisoning and procedural complications) | 1 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 2
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase (Investigations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 15 | 3
Amylase increased (Investigations) | 1 | 0
Aspartate aminotransferase (Investigations) | 0 | 1
Erythropenia (Blood and lymphatic system disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 175 | 65
Peritonsillitis (Infections and infestations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 16 | 2
Basophil count increased (Investigations) | 1 | 0
Blood albumin decreased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 3 | 1
Blood bicarbonate increased (Investigations) | 3 | 2
Blood bilirubin increased (Investigations) | 4 | 1
Blood calcium decreased (Investigations) | 1 | 0
Blood chloride decreased (Investigations) | 0 | 1
Blood chloride increased (Investigations) | 0 | 1
Blood cholesterol increased (Investigations) | 1 | 0
Blood creatine abnormal (Investigations) | 0 | 1
Blood creatine increased (Investigations) | 1 | 0
Blood creatine phosphokinase MB increased (Investigations) | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 17 | 18
Blood creatinine increased (Investigations) | 21 | 24
Blood glucose increased (Investigations) | 4 | 2
Blood lactate dehydrogenase decreased (Investigations) | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 15 | 3
Blood magnesium decreased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 1 | 0
Blood potassium increased (Investigations) | 0 | 3
Blood pressure diastolic increased (Investigations) | 1 | 2
Blood pressure increased (Investigations) | 6 | 2
Blood pressure orthostatic (Investigations) | 1 | 0
Blood pressure systolic increased (Investigations) | 1 | 3
Blood sodium decreased (Investigations) | 0 | 1
Blood thyroid stimulating hormone decreased (Investigations) | 6 | 1
Blood thyroid stimulating hormone increased (Investigations) | 23 | 7
Blood triglycerides increased (Investigations) | 0 | 1
Blood urea increased (Investigations) | 5 | 7
Blood uric acid increased (Investigations) | 3 | 2
Body temperature increased (Investigations) | 1 | 0
Cardiac murmur (Investigations) | 0 | 2
Cardiac stress test abnormal (Investigations) | 1 | 0
Chest X-ray abnormal (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 3 | 6
Electrocardiogram QT interval abnormal (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 4 | 1
Electrocardiogram ST segment abnormal (Investigations) | 1 | 0
Electrocardiogram ST segment depression (Investigations) | 1 | 0
Electrocardiogram ST segment elevation (Investigations) | 0 | 1
Electrocardiogram ST-T change (Investigations) | 1 | 2
Electrocardiogram T wave inversion (Investigations) | 1 | 0
Electrocardiogram T wave peaked (Investigations) | 1 | 0
Eosinophil count increased (Investigations) | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 2 | 1
Haemoglobin decreased (Investigations) | 9 | 2
Hepatic enzyme increased (Investigations) | 2 | 2
International normalised ratio increased (Investigations) | 1 | 0
Liver function test increased (Investigations) | 1 | 0
Low density lipoprotein increased (Investigations) | 1 | 0
Monocyte count increased (Investigations) | 1 | 0
Neutrophil count (Investigations) | 2 | 0
Neutrophil count decreased (Investigations) | 13 | 3
Platelet count (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 8 | 1
Platelet count increased (Investigations) | 0 | 2
Prostatic specific antigen increased (Investigations) | 1 | 2
Protein total decreased (Investigations) | 3 | 0
Protein total increased (Investigations) | 1 | 2
Protein urine present (Investigations) | 2 | 0
QRS axis abnormal (Investigations) | 1 | 0
Red blood cell count increased (Investigations) | 0 | 1
Staphylococcus test positive (Investigations) | 1 | 0
Thyroid function test abnormal (Investigations) | 1 | 0
Thyroxine decreased (Investigations) | 1 | 0
Thyroxine free decreased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 2 | 0
Troponin T increased (Investigations) | 1 | 0
Visual acuity tests (Investigations) | 1 | 0
Weight decreased (Investigations) | 14 | 2
Weight increased (Investigations) | 8 | 18
White blood cell count (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 15 | 2
Xanthochromia (Investigations) | 1 | 0
Alkalosis (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 59 | 16
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 4 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 7
Hypercreatininaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 11
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 1
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 7 | 3
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0
Hypovitaminosis (Metabolism and nutrition disorders) | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 35 | 29
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 28 | 26
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 8
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 2
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Groin pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Interspinous osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 4 | 2
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 25 | 13
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 13 | 14
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 25 | 15
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 5
Nodal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 3
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis postmenopausal (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 45 | 20
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Spinal pain (Musculoskeletal and connective tissue disorders) | 8 | 2
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Ageusia (Nervous system disorders) | 21 | 0
Aphonia (Nervous system disorders) | 1 | 1
Balance disorder (Nervous system disorders) | 0 | 1
Burning sensation (Nervous system disorders) | 1 | 0
Carotid arteriosclerosis (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Disturbance in attention (Nervous system disorders) | 2 | 1
Dizziness (Nervous system disorders) | 23 | 18
Dizziness postural (Nervous system disorders) | 1 | 0
Dysaesthesia (Nervous system disorders) | 4 | 1
Dysgeusia (Nervous system disorders) | 103 | 18
Facial nerve disorder (Nervous system disorders) | 1 | 0
Facial paralysis (Nervous system disorders) | 0 | 1
Formication (Nervous system disorders) | 0 | 2
Head discomfort (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 56 | 36
Hyperaesthesia (Nervous system disorders) | 5 | 3
Hypoaesthesia (Nervous system disorders) | 4 | 1
Hypogeusia (Nervous system disorders) | 2 | 0
Hypotonia (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 9 | 9
Loss of consciousness (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 4 | 3
Migraine (Nervous system disorders) | 2 | 0
Muscle contractions involuntary (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 7 | 4
Paraesthesia (Nervous system disorders) | 12 | 11
Parkinson's disease (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 7
Polyneuropathy (Nervous system disorders) | 1 | 1
Presyncope (Nervous system disorders) | 1 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 1
Sciatica (Nervous system disorders) | 6 | 0
Seizure (Nervous system disorders) | 1 | 0
Sensory disturbance (Nervous system disorders) | 2 | 0
Sensory loss (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Tongue paralysis (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 3 | 3
Affective disorder (Psychiatric disorders) | 1 | 2
Agitated depression (Psychiatric disorders) | 0 | 1
Agitation (Psychiatric disorders) | 1 | 0
Anger (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 10 | 14
Apathy (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Depressed mood (Psychiatric disorders) | 3 | 4
Depression (Psychiatric disorders) | 3 | 10
Insomnia (Psychiatric disorders) | 30 | 19
Irritability (Psychiatric disorders) | 5 | 4
Listless (Psychiatric disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 0 | 1
Mood altered (Psychiatric disorders) | 5 | 3
Nervousness (Psychiatric disorders) | 4 | 2
Persecutory delusion (Psychiatric disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 3 | 1
Stress (Psychiatric disorders) | 1 | 0
Tension (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Albuminuria (Renal and urinary disorders) | 0 | 1
Bladder disorder (Renal and urinary disorders) | 0 | 1
Bladder pain (Renal and urinary disorders) | 0 | 1
Bladder spasm (Renal and urinary disorders) | 0 | 1
Chromaturia (Renal and urinary disorders) | 9 | 0
Dysuria (Renal and urinary disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 7 | 5
Nocturia (Renal and urinary disorders) | 1 | 6
Pollakiuria (Renal and urinary disorders) | 0 | 3
Proteinuria (Renal and urinary disorders) | 18 | 9
Pyelocaliectasis (Renal and urinary disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 1
Renal impairment (Renal and urinary disorders) | 1 | 2
Renal pain (Renal and urinary disorders) | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Amenorrhoea (Reproductive system and breast disorders) | 1 | 0
Balanoposthitis (Reproductive system and breast disorders) | 2 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 3
Breast engorgement (Reproductive system and breast disorders) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 2 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 2 | 0
Genital rash (Reproductive system and breast disorders) | 2 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 3
Haematospermia (Reproductive system and breast disorders) | 1 | 0
Breast tenderness (Reproductive system and breast disorders) | 0 | 1
Menometrorrhagia (Reproductive system and breast disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 2 | 0
Ovarian disorder (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 2 | 2
Penile pain (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1
Scrotal erythema (Reproductive system and breast disorders) | 1 | 0
Scrotal pain (Reproductive system and breast disorders) | 2 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 3
Testicular swelling (Reproductive system and breast disorders) | 1 | 0
Testis discomfort (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 22 | 20
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 10 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 | 19
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 55 | 9
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 17 | 10
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 6 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 26 | 2
Blister (Skin and subcutaneous tissue disorders) | 6 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 5 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 43 | 17
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 5 | 3
Erythema (Skin and subcutaneous tissue disorders) | 13 | 10
Erythrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 5 | 0
Granuloma annulare (Skin and subcutaneous tissue disorders) | 1 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 68 | 7
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 2 | 0
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 2
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 10 | 2
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0
Keloid scar (Skin and subcutaneous tissue disorders) | 0 | 1
Macule (Skin and subcutaneous tissue disorders) | 1 | 0
Nail bed bleeding (Skin and subcutaneous tissue disorders) | 1 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 6 | 2
Nail growth abnormal (Skin and subcutaneous tissue disorders) | 2 | 0
Nail toxicity (Skin and subcutaneous tissue disorders) | 3 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 2
Palmar erythema (Skin and subcutaneous tissue disorders) | 2 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 154 | 31
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 5 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 3 | 2
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 2 | 0
Plantar erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 21 | 21
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 59 | 29
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 2
Rash follicular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 2 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 4 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 | 0
Scar pain (Skin and subcutaneous tissue disorders) | 1 | 7
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 | 1
Skin depigmentation (Skin and subcutaneous tissue disorders) | 2 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 24 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 11 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 3 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 12 | 2
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 9 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 9 | 2
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 1
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 1 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 2 | 0
Splinter haemorrhages (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 5 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 1
Urticaria thermal (Skin and subcutaneous tissue disorders) | 0 | 1
Yellow skin (Skin and subcutaneous tissue disorders) | 33 | 2
Disability (Social circumstances) | 1 | 0
Walking disability (Social circumstances) | 1 | 0
Abdominal hernia repair (Surgical and medical procedures) | 1 | 0
Cancer surgery (Surgical and medical procedures) | 1 | 0
Hysterectomy (Surgical and medical procedures) | 1 | 0
Injection (Surgical and medical procedures) | 1 | 0
Palatal operation (Surgical and medical procedures) | 1 | 0
Spleen operation (Surgical and medical procedures) | 1 | 0
Therapeutic procedure (Surgical and medical procedures) | 1 | 0
Tooth extraction (Surgical and medical procedures) | 2 | 1
Wisdom teeth removal (Surgical and medical procedures) | 1 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1
Capillary disorder (Vascular disorders) | 1 | 0
Embolism venous (Vascular disorders) | 1 | 0
Endothelial dysfunction (Vascular disorders) | 1 | 0
Flushing (Vascular disorders) | 3 | 1
Haematoma (Vascular disorders) | 3 | 1
Hot flush (Vascular disorders) | 4 | 3
Hypertension (Vascular disorders) | 112 | 35
Hypertensive crisis (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 4 | 3
Infarction (Vascular disorders) | 1 | 0
Pallor (Vascular disorders) | 1 | 1
Peripheral coldness (Vascular disorders) | 2 | 1
Phlebitis (Vascular disorders) | 1 | 1
Phlebolith (Vascular disorders) | 0 | 1
Poor peripheral circulation (Vascular disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7 | 4
Dental implantation (Surgical and medical procedures) | 0 | 1
Gingival discomfort (Gastrointestinal disorders) | 1 | 0
Tongue discomfort (Gastrointestinal disorders) | 3 | 0
Sensation of foreign body (General disorders) | 1 | 0
Urobilinogen urine increased (Investigations) | 1 | 0
Irregular sleep wake rhythm disorder (Nervous system disorders) | 1 | 0
Red blood cell count decreased (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.